CLINICAL TRIAL: NCT03627494
Title: A Three-Part FTIH Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Repeat Oral Doses of GSK3439171A, in a Randomized, Double-Blind (Sponsor Unblinded), Placebo-Controlled, Dose Escalation Study and to Evaluate the Effect of Food on a Single Oral Dose of GSK3439171A in Healthy Adult Participants
Brief Title: First Time in Human (FTIH) Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Single and Repeat Doses of GSK3439171A in Healthy Subjects and to Assess Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 209275
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Results first posted 2020-07-10 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-05

CONDITIONS: Muscular Dystrophies
Keywords: Dose proportionality; Food effect; Pharmacokinetics; FTIH; Pharmacodynamics; Dose Escalation
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: Part A is a Crossover group single ascending dose study with 2 arms per cohort that is subject and investigator blinded. Part B is a Parallel group repeat dose study with 2 arms per cohort that is subject and investigator blinded. Part C is a Crossover group food effect study with 2 arms per cohort that is not-masked."
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part A: P1,PBO/GSK3439171A Dose 2/GSK3439171A Dose 3 (Experimental): Subjects will administer oral solution with doses 0.5 milligram (mg) up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A and placebo as per randomized sequence placebo (PBO) followed by Dose 2 of GSK3439171A followed by Dose 3 of GSK3439171A in period 1 (P1). There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part A: P1, GSK3439171A Dose 1/ PBO/GSK3439171A Dose 3 (Experimental): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A and PBO as per randomized sequence: Dose 1 of GSK3439171A followed by PBO followed by Dose 3 of GSK3439171A in P1. There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part A: P1, GSK3439171A Dose 1/ GSK3439171A Dose 2/ PBO (Experimental): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A and placebo as per randomized sequence: Dose 1 of GSK3439171A followed by Dose 2 of GSK3439171A followed by PBO in P1. There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part A: P2, PBO/GSK3439171A Dose 5/GSK3439171A Dose 6 (Experimental): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A and placebo as per randomized sequence: PBO followed by Dose 5 of GSK3439171A followed by Dose 6 of GSK3439171A in period 2 (P2). There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part A: P2, GSK3439171A Dose 4/ PBO/GSK3439171A Dose 6 (Experimental): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A and placebo as per randomized sequence: Dose 4 of GSK3439171A followed by PBO followed by Dose 6 of GSK3439171A in P2. There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part A: P2, GSK3439171A Dose 4/ GSK3439171A Dose 5/ PBO (Experimental): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A and placebo as per randomized sequence: Dose 4 of GSK3439171A followed by Dose 5 of GSK3439171A followed by PBO in P2. There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part A: P3, PBO/GSK3439171A Dose 8/GSK3439171A Dose 9 (Experimental): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A and placebo as per randomized sequence: PBO followed by Dose 8 of GSK3439171A followed by Dose 9 of GSK3439171A in Period 3 (P3). There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part A: P3, GSK3439171A Dose 7/ PBO/GSK3439171A Dose 9 (Experimental): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A and placebo as per randomized sequence: Dose 7 of GSK3439171A followed by PBO followed by Dose 9 of GSK3439171A in P3. There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part A: P3, GSK3439171A Dose 7/ GSK3439171A Dose 8/ PBO (Experimental): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A and placebo as per randomized sequence: Dose 7 of GSK3439171A followed by Dose 8 of GSK3439171A followed by PBO in P3. There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part B: GSK3439171A (Experimental): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of GSK3439171A in part B
  Interventions: Drug: GSK3439171A
- Part B: Placebo (Placebo Comparator): Subjects will administer oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards of Placebo in part B
  Interventions: Drug: Placebo
- Part C: GSK3439171A fed followed by GSK3439171A fasted (Experimental): Subjects will administer GSK3439171A in Fed condition in Part C P1 followed by GSK3439171A in fasted condition in Part C P2. There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo
- Part C: GSK3439171A fasted followed by GSK3439171A fed (Experimental): Subjects will administer GSK3439171A in fasted condition in Part C P1 followed by GSK3439171A in fed condition in Part C P2. There will be a washout period of 7 days or 5 half-lives, whichever is longer in between the doses.
  Interventions: Drug: GSK3439171A; Drug: Placebo

INTERVENTIONS:
Drug: GSK3439171A — Oral solution with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards
  Arms: Part A: P1, GSK3439171A Dose 1/ GSK3439171A Dose 2/ PBO; Part A: P1, GSK3439171A Dose 1/ PBO/GSK3439171A Dose 3; Part A: P1,PBO/GSK3439171A Dose 2/GSK3439171A Dose 3; Part A: P2, GSK3439171A Dose 4/ GSK3439171A Dose 5/ PBO; Part A: P2, GSK3439171A Dose 4/ PBO/GSK3439171A Dose 6; Part A: P2, PBO/GSK3439171A Dose 5/GSK3439171A Dose 6; Part A: P3, GSK3439171A Dose 7/ GSK3439171A Dose 8/ PBO; Part A: P3, GSK3439171A Dose 7/ PBO/GSK3439171A Dose 9; Part A: P3, PBO/GSK3439171A Dose 8/GSK3439171A Dose 9; Part B: GSK3439171A; Part C: GSK3439171A fasted followed by GSK3439171A fed; Part C: GSK3439171A fed followed by GSK3439171A fasted
Drug: Placebo — Placebo oral solution to match with doses 0.5 mg up to 4.5 mg and capsule for doses 5 mg and upwards
  Arms: Part A: P1, GSK3439171A Dose 1/ GSK3439171A Dose 2/ PBO; Part A: P1, GSK3439171A Dose 1/ PBO/GSK3439171A Dose 3; Part A: P1,PBO/GSK3439171A Dose 2/GSK3439171A Dose 3; Part A: P2, GSK3439171A Dose 4/ GSK3439171A Dose 5/ PBO; Part A: P2, GSK3439171A Dose 4/ PBO/GSK3439171A Dose 6; Part A: P2, PBO/GSK3439171A Dose 5/GSK3439171A Dose 6; Part A: P3, GSK3439171A Dose 7/ GSK3439171A Dose 8/ PBO; Part A: P3, GSK3439171A Dose 7/ PBO/GSK3439171A Dose 9; Part A: P3, PBO/GSK3439171A Dose 8/GSK3439171A Dose 9; Part B: Placebo; Part C: GSK3439171A fasted followed by GSK3439171A fed; Part C: GSK3439171A fed followed by GSK3439171A fasted

SUMMARY:
The FTIH study with GSK3439171A will evaluate the safety of GSK3439171A in healthy subjects in order to avoid confounding factors due to the disease or concomitant drugs in patients. The study design is based on pre-clinical findings for GSK3439171A, contributing to the frequency, type and duration of safety assessment and monitoring during treatment periods in each cohort. The single dose assessments in Part A will be conducted to determine safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of the study intervention in individuals before progressing to doses explored further in other parts of the study and will allow for any adjustments needed based on emerging safety, tolerability, and PK information. Part A will also serve to identify a dose for use in examining the effect of food on GSK3439171A exposure in Part C. In Part B, a single dose safety, tolerability and PK will be collected followed by progression of these subjects to the repeat dose portion of the study. The up to 14-day dosing was chosen as it is thought to provide sufficient safety and tolerability data to bridge to longer duration studies. The dosing period can be adjusted depending on PK and PD data collected in Part A of the study. Part B will involve more detailed PK/PD/metabolite assessments to better understand the impact of GSK3439171A on target engagement and metabolism in humans. Approximately 150 subjects will be screened to achieve 75 randomly assigned to study intervention. Duration for Part A, B and C will be approximately 10 weeks, 9 weeks and 8 weeks respectively.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 to 65 years of age inclusive, at the time of signing the informed consent.
* Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) not specifically listed in the exclusion or exclusion criteria that is outside the reference range for the population being studied may be included only if the investigator, in consultation with the Medical Monitor, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subjects with Body weight >=50.0 kilograms (Kg) (110 lbs.) and body mass index (BMI) within the range 18.5 to 31.0 kilograms per square meter (inclusive).
* Only male subjects are eligible for this study. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male subjects are eligible to participate if they agree to the following during the their entire enrolment in the study plus an additional 5 days or 5 terminal half-lives (whichever is longer): Refrain from donating sperm plus either be abstinent from sexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or must agree to use contraception/barrier (female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year)
* Subjects must be capable of giving signed informed consent

Exclusion Criteria:

* Subjects are excluded from the study if they have history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Subjects are excluded from the study if they have any clinically significant abnormal vital signs
* Subjects are excluded from the study if they have Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Subjects are excluded from the study if they have ALT >1.5 times upper limit of normal (ULN)
* Subjects are excluded from the study if Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Subjects are excluded from the study if they have current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects are excluded from the study if they have QTc >450 milliseconds
* Subjects who are unable to refrain from the use of prescription or non-prescription drugs, including aspirin, Non-steroidal Anti-inflammatory Drugs (NSAIDs), vitamins, herbal and dietary supplements (including St John's Wort) within 10 days prior to the first dose of study medication.
* In cases, where participation in the study would result in loss of blood or blood products in excess of 500 milliliter (mL) within 56 days
* Subjects with exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Subjects with current enrolment or past participation within the last 30 days before signing of consent in this or any other clinical study involving an investigational study intervention or any other type of medical research.
* Subjects with presence of Hepatitis B surface antigen (HBsAg) at screening.
* Subjects with Positive Hepatitis C antibody test result at screening. Subjects with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C ribonucleic acid (RNA) test is obtained.
* Subjects with Positive Hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention
* Subjects with positive pre-study drug/alcohol screen
* Subjects with positive human immunodeficiency virus (HIV) antibody test
* Subjects with regular use of known drugs of abuse or positive urine drug test at screening or each in-house admission to the clinical research unit
* Subjects with regular alcohol consumption within 6 months prior to screening and 5 days prior to admission defined as: An average weekly intake of > 14 units for males. One unit is equivalent to 8 gram of alcohol: a half-pint (Approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of 80 proof distilled spirits
* Subjects with positive urinary cotinine test indicative of smoking history at screening or each in-house admission to the clinical research unit or regular use of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) within 6 months prior to screening
* Subjects with sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males are eligible for this study
Enrollment: 66 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request Site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 3 part study conducted at a single center in the United States where, Part A is a single oral dose, dose-rising, 3 period crossover study; Part B is a repeat oral dosing, dose escalation study and Part C is a crossover study where a single dose was administered in fasted or fed conditions.
Pre-assignment Details: A total of 66 participants were enrolled in Part A (18 participants), Part B (36 participants) and Part C (12 participants).
Groups:
- GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg: Participants were administered a single oral dose of 5 milligrams (mg) GSK3439171A on Day 1 of treatment period 1, followed by a single oral dose of placebo on Day 1 of treatment period 2. Participants were further administered a single oral dose of 30 mg GSK3439171A on Day 1 of treatment period 3. There was a washout of 7 days between dosing in each treatment period. All participants were followed up for 14 days after the administration of last dose of study treatment.
- Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg: Participants were administered a single oral dose of placebo on Day 1 of treatment period 1 followed by a single oral dose of 10 mg GSK3439171A on Day 1 of treatment period 2. Participants were further administered a single oral dose of 30 mg GSK3439171A in treatment period 3. There was a washout of 7 days between dosing in each treatment period. All participants were followed up for 14 days after the administration of last dose of study treatment.
- GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo: Participants were administered a single oral dose of 5 mg GSK3439171A on Day 1 of treatment period 1 followed by a single oral dose of 10 mg GSK3439171A on Day 1 of treatment period 2. Participants were further administered a single oral dose of placebo on Day 1 of treatment period 3. There was a washout of 7 days between dosing in each treatment period. All participants were followed up for 14 days after the administration of last dose of study treatment.
- GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo: Participants were administered a single oral dose of 60 mg GSK3439171A on Day 1 of treatment period 1 followed by a single oral dose of 120 mg GSK3439171A on Day 1 of treatment period 2. Participants then administered a single oral dose of placebo on Day 1 of treatment period 3. There was a washout of 7 days between dosing in each treatment period. All participants were followed up for 14 days after the administration of last dose of study treatment.
- Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg: Participants were administered a single oral dose of placebo on Day 1 of treatment period 1 followed by a single oral dose of 120 mg GSK3439171A on Day 1 of treatment period 2. Participants were further administered a single oral dose of 180 mg GSK3439171A on Day 1 of treatment period 3. There was a washout of 7 days between dosing in each treatment period. All participants were followed up for 14 days after the administration of last dose of study treatment.
- GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg: Participants were administered a single oral dose of 60 mg GSK3439171A on Day 1 of treatment period 1 followed by a single oral dose of placebo on Day 1 of treatment period 2. Participants were further administered a single oral dose of 180 mg GSK3439171A on Day 1 of treatment period 3. There was a washout of 7 days between dosing in each treatment period. All participants were followed up for 14 days after the administration of last dose of study treatment.
- Placebo: Participants were administered placebo once daily via oral route for 13 or 20 days. All participants were followed up for 14 days after the administration of last dose of study treatment.
- GSK3439171A 5 mg: Participants were administered GSK343917A 5 mg once daily via oral route for 20 days. All participants were followed up for 14 days after the administration of last dose of study treatment.
- GSK3439171A 11 mg: Participants were administered GSK343917A 11 mg once daily via oral route for 20 days. All participants were followed up for 14 days after the administration of last dose of study treatment.
- GSK3439171A 40 mg: Participants were administered GSK343917A 40 mg once daily via oral route for 13 days. All participants were followed up for 14 days after the administration of last dose of study treatment.
- GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed: Participants were administered a single oral dose of GSK3439171A 60 mg in the fasted state on Day 1 of treatment period 1 followed by a washout of 7 days. In treatment period 2, participants were administered a single oral dose of GSK3439171A 60 mg after a high fat meal. All participants were followed up for 14 days after the administration of last dose of study treatment.
- GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted: Participants were administered a single oral dose of GSK3439171A 60 mg after a high fat meal on Day 1 of treatment period 1 followed by a washout of 7 days. In treatment period 2, participants were administered a single oral dose of GSK3439171A 60 mg in the fasted state. All participants were followed up for 14 days after the administration of last dose of study treatment.
Period: Part A Period 1 (4 Days)
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed (0) | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Washout 1 (7 Days)
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period 2 (4 Days)
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Washout 2 (7 Days)
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Period3(4days)+Follow-up(14days)
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted
Started | 2 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Maximum of 34 Days)
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted
Started | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 9 | 9 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 7 | 9 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Period: Part C Period 1 (4 Days)
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C Washout 1 (7 Days)
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Period: Part C Period2(4days)+Follow-up(14days)
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3439171A 5 mg/Placebo/GSK3439171A 30 mg | Placebo/ GSK3439171A 10 mg/GSK3439171A 30 mg | GSK3439171A 5 mg/GSK3439171A 10 mg/Placebo | GSK3439171A 60 mg/GSK3439171A 120 mg/Placebo | Placebo/ GSK3439171A 120 mg/GSK3439171A 180 mg | GSK3439171A 60 mg/Placebo/GSK3439171A 180 mg | Placebo | GSK3439171A 5 mg | GSK3439171A 11 mg | GSK3439171A 40 mg | GSK3439171A 60 mg Fasted/GSK3439171A 60 mg Fed | GSK3439171A 60 mg Fed/GSK3439171A 60 mg Fasted | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 9 | 9 | 9 | 6 | 6 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (4.58) | 43.0 (2.65) | 37.3 (11.85) | 44.3 (12.50) | 49.0 (9.17) | 42.0 (7.55) | 46.7 (8.83) | 37.6 (9.26) | 45.0 (8.80) | 41.6 (10.31) | 38.3 (12.89) | 47.8 (6.21) | 42.7 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 9 | 9 | 9 | 6 | 6 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-East Asian Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Black or African American | 1 | 3 | 3 | 2 | 1 | 2 | 3 | 3 | 4 | 3 | 2 | 4 | 31
  White-White/Caucasian/European Heritage | 2 | 0 | 0 | 1 | 2 | 1 | 5 | 5 | 5 | 6 | 3 | 2 | 32
  Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)-Part A
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; other important medical events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed before.
Time Frame: Up to Day 40
Population: Safety Population comprised of all participants who took at least one dose of study intervention. Participants were analyzed according to the intervention they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Placebo: Participants were administered a single oral dose of placebo on Day 1 of treatment period 1, 2 or 3.
- Part A: GSK3439171A 5 mg: Participants were administered a single oral dose of GSK3439171A 5 mg on Day 1 of either treatment period 1, 2 or 3.
- Part A: GSK3439171A 10 mg: Participants were administered a single oral dose of GSK3439171A 10 mg on Day 1 of either treatment period 1, 2 or 3.
- Part A: GSK3439171A 30 mg: Participants were administered a single oral dose of GSK3439171A 30 mg on Day 1 of either treatment period 1, 2 or 3.
- Part A: GSK3439171A 60 mg: Participants were administered a single oral dose of GSK3439171A 60 mg on Day 1 of either treatment period 1, 2 or 3.
- Part A: GSK3439171A 120 mg: Participants were administered a single oral dose of GSK3439171A 120 mg on Day 1 of either treatment period 1, 2 or 3.
- Part A: GSK3439171A 180 mg: Participants were administered a single oral dose of GSK3439171A 180 mg on Day 1 of either treatment period 1, 2 or 3.
Arm/Group | Part A: Placebo | Part A: GSK3439171A 5 mg | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 17 | 6 | 6 | 5 | 6 | 6 | 6
Participants
  Any AE | 1 | 0 | 2 | 2 | 2 | 1 | 1
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With AEs and SAEs-Part B
Description: as for outcome 1
Time Frame: Up to Day 34
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Placebo: Participants were administered placebo once daily via oral route for 13 or 20 days. All participants were followed up for 14 days after the administration of last dose of study treatment.
- Part B: GSK3439171A 5 mg: Participants were administered GSK343917A 5 mg once daily via oral route for 20 days. All participants were followed up for 14 days after the administration of last dose of study treatment.
- Part B: GSK3439171A 11 mg: Participants were administered GSK343917A 11 mg once daily via oral route for 20 days. All participants were followed up for 14 days after the administration of last dose of study treatment.
- Part B: GSK3439171A 40 mg: Participants were administered GSK343917A 40 mg once daily via oral route for 13 days. All participants were followed up for 14 days after the administration of last dose of study treatment.
Arm/Group | Part B: Placebo | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Any AE | 4 | 5 | 8 | 3
  Any SAE | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With AEs and SAEs-Part C
Description: as for outcome 1
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part C: GSK3439171A 60 mg Fasted: Participants were administered a single oral dose of GSK3439171A 60 mg in the fasted state on Day 1 of either treatment period 1 or 2.
- Part C: GSK3439171A 60 mg Fed: Participants were administered a single oral dose of GSK3439171A 60 mg after a high fat meal on Day 1 of either treatment period 1 or 2.
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Participants
  Any AE | 1 | 3
  Any SAE | 0 | 0

4. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance-Part A
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The clinical concern range for the parameters were: albumin (low: <30 grams per liter [g/L]); alanine aminotransferase (ALT) (high: >=2xupper limit of normal [ULN]); aspartate aminotransferase (AST) (high: >=2xULN); alkaline phosphatase (ALP) (high: >=2xULN); total bilirubin (high: >=1.5xULN); calcium (low: <2 millimoles (mmol)/L and high: >2.75 mmol/L); creatinine (high: change from Baseline >44.2 micromoles/L); glucose (low: <3 mmol/L and high: >9 mmol/L); magnesium (low: 0.5 mmol/L and high: 1.23 mmol/L); phosphorus (low: 0.8 mmol/L and high: 1.6 mmol/L); potassium (low: <3 mmol/L and high: >5.5 mmol/L); sodium (low: <130 mmol/L and high: >150 mmol/L) and creatine kinase (high: >500 units per liter). The number of participants with any clinical chemistry abnormality of potential clinical importance is reported.
Time Frame: Up to Day 40
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3439171A 5 mg | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 17 | 6 | 6 | 5 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 1

5. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance-Part B
Description: Blood samples were collected for the assessment of clinical chemistry parameters. The clinical concern range for the parameters were: albumin (low: <30 g/L); ALT (high: >=2xULN); AST (high: >=2xULN); ALP (high: >=2xULN); total bilirubin (high: >=1.5xULN); calcium (low: <2 mmol/L and high: >2.75 mmol/L); creatinine (high: change from Baseline >44.2 micromoles/L); glucose (low: <3 mmol/L and high: >9 mmol/L); magnesium (low: 0.5 mmol/L and high: 1.23 mmol/L); phosphorus (low: 0.8 mmol/L and high: 1.6 mmol/L); potassium (low: <3 mmol/L and high: >5.5 mmol/L); sodium (low: <130 mmol/L and high: >150 mmol/L) and creatine kinase (high: >500 units per liter). The number of participants with any clinical chemistry abnormality of potential clinical importance is reported.
Time Frame: Up to Day 34
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 1

6. Primary Outcome: Number of Participants With Clinical Chemistry Abnormalities of Potential Clinical Importance-Part C
Description: as for outcome 5
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Participants | 0 | 0

7. Primary Outcome: Number of Participants With Hematology Abnormalities of Potential Clinical Importance-Part A
Description: Blood samples were collected for the assessment of hematology parameters. The clinical concern range for the parameters were: hematocrit (high: >0.54 proportion of red blood cells in blood); hemoglobin (high: >180 g/L), lymphocytes (low: <0.8x10^9 cells per liter [cells/L]); neutrophil count (low: <1.5x10^9 cells/L); platelet count (low: <100x10^9 cells/L and high: >550x10^9 cells/L); white blood cells count (low: <3x10^9 cells/L and high: >20x10^9 cells/L). The number of participants with any hematology abnormality of potential clinical importance is reported.
Time Frame: Up to Day 40
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3439171A 5 mg | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 17 | 6 | 6 | 5 | 6 | 6 | 6
Participants | 2 | 0 | 1 | 0 | 1 | 1 | 1

8. Primary Outcome: Number of Participants With Hematology Abnormalities of Potential Clinical Importance-Part B
Description: Blood samples were collected for the assessment of hematology parameters. The clinical concern range for the parameters were: hematocrit (high: >0.54 proportion of red blood cells in blood); hemoglobin (high: >180 g/L), lymphocytes (low: <0.8x10^9 cells/L); neutrophil count (low: <1.5x10^9 cells/L); platelet count (low: <100x10^9 cells/L and high: >550x10^9 cells/L); white blood cells count (low: <3x10^9 cells/L and high: >20x10^9 cells/L). The number of participants with any hematology abnormality of potential clinical importance is reported.
Time Frame: Up to Day 34
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 3 | 3 | 2 | 1

9. Primary Outcome: Number of Participants With Hematology Abnormalities of Potential Clinical Importance-Part C
Description: as for outcome 8
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Participants | 5 | 3

10. Primary Outcome: Number of Participants With Abnormal Urinalysis Dipstick Results-Part A
Description: Urine samples were taken for the assessment of following urine parameters: glucose, ketones, occult blood (OB) and protein by dipstick method. The dipstick test gives results in a semi-quantitative manner, and results can be read as Trace, 1+, 2+ indicating proportional concentrations in the urine sample.
Time Frame: 8 hours, 24 hours, 48 hours and 72 hours in Periods 1, 2 and 3
Population: Safety Population. All participants in Part A (17, 6, 6, 5, 6, 6, 6) were included in the analysis; however, only participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3439171A 5 mg | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 17 | 6 | 6 | 5 | 6 | 6 | 6
Participants
  Glucose; Period 1; 8 hours;Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 8 hours;Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Glucose; Period 1; 8 hours;1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 8 hours;1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Glucose; Period 1; 8 hours;2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 8 hours;2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Glucose; Period 1; 24 hours;Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 24 hours;Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Glucose; Period 1; 24 hours;1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 24 hours;1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Glucose; Period 1; 24 hours;2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 24 hours;2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Glucose; Period 1; 48 hours;Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 48 hours;Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Glucose; Period 1; 48 hours;1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 48 hours;1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Glucose; Period 1; 48 hours;2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 48 hours;2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Glucose; Period 1; 72 hours;Trace;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 72 hours;Trace;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Glucose; Period 1; 72 hours;1+;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 72 hours;1+;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Glucose; Period 1; 72 hours;2+;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Glucose; Period 1; 72 hours;2+;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Glucose; Period 2; 8 hours;Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 8 hours;Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  | 0 | 0 |
  Glucose; Period 2; 8 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 8 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 8 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 8 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 24 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 24 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 24 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 24 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 24 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 24 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 48 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 48 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 48 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 48 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 48 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 48 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 72 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 72 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 72 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 72 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 2; 72 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Glucose; Period 2; 72 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Glucose; Period 3; 8 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 8 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 8 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 8 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 8 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 8 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 24 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 24 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 24 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 24 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 24 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 24 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 48 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 48 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 48 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 48 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 48 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 48 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 72 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 72 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 72 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 72 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Glucose; Period 3; 72 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Glucose; Period 3; 72 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 1; 8 hours; Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 8 hours; Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Ketones; Period 1; 8 hours; 1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 8 hours; 1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Ketones; Period 1; 8 hours; 2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 8 hours; 2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Ketones; Period 1; 24 hours; Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 24 hours; Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Ketones; Period 1; 24 hours; 1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 24 hours; 1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Ketones; Period 1; 24 hours;2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 24 hours;2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Ketones; Period 1; 48 hours; Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 48 hours; Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Ketones; Period 1; 48 hours; 1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 48 hours; 1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Ketones; Period 1; 48 hours; 2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 48 hours; 2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Ketones; Period 1; 72 hours; Trace;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 72 hours; Trace;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Ketones; Period 1; 72 hours; 1+;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 72 hours; 1+;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Ketones; Period 1; 72 hours; 2+;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Ketones; Period 1; 72 hours; 2+;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Ketones; Period 2; 8 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 8 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 8 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 8 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 8 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 8 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 24 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 24 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 24 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 24 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 24 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 24 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 48 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 48 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 00 |
  Ketones; Period 2; 48 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 48 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 48 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 48 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 72 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 72 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 72 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 72 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 2; 72 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Ketones; Period 2; 72 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Ketones; Period 3; 8 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 8 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 8 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 8 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 8 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 8 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 24 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 24 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 24 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 24 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 24 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 24 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 48 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 48 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 48 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 48 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 72 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 72 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 72 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 72 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Ketones; Period 3; 72 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Ketones; Period 3; 72 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 1; 8 hours; Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 8 hours; Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  OB; Period 1; 8 hours; 1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 8 hours; 1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  OB; Period 1; 8 hours; 2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 8 hours; 2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  OB; Period 1; 24 hours; Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 24 hours; Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  OB; Period 1; 24 hours; 1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 24 hours; 1+;n=6,6,0,0,6,0,0 | 1 | 0 |  |  | 0 |  |
  OB; Period 1; 24 hours;2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 24 hours;2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  OB; Period 1; 48 hours; Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 48 hours; Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  OB; Period 1; 48 hours; 1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 48 hours; 1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  OB; Period 1; 48 hours; 2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 48 hours; 2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  OB; Period 1; 72 hours; Trace;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 72 hours; Trace;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  OB; Period 1; 72 hours; 1+;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 72 hours; 1+;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  OB; Period 1; 72 hours; 2+;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  OB; Period 1; 72 hours; 2+;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  OB; Period 2; 8 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 8 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  OB; Period 2; 8 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 8 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 1 |
  OB; Period 2; 8 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 8 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  OB; Period 2; 24 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 24 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  OB; Period 2; 24 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 24 hours; 1+;n=6,0,6,0,0,6,0 | 1 |  | 1 |  |  | 1 |
  OB; Period 2; 24 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 24 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  OB; Period 2; 48 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 48 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  OB; Period 2; 48 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 48 hours; 1+;n=6,0,6,0,0,6,0 | 1 |  | 0 |  |  | 0 |
  OB; Period 2; 48 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 48 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  OB; Period 2; 72 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 72 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  OB; Period 2; 72 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 72 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 1 |
  OB; Period 2; 72 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  OB; Period 2; 72 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  OB; Period 3; 8 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 8 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 3; 8 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 8 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 1 |  |  | 0
  OB; Period 3; 8 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 8 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 3; 24 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 24 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 3; 24 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 24 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 3; 24 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 24 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 3; 48 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 48 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 3; 48 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 48 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 3; 48 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 48 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 3; 72 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 72 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  OB; Period 3; 72 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 72 hours; 1+;n=5,0,0,5,0,0,6 | 1 |  |  | 0 |  |  | 2
  OB; Period 3; 72 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  OB; Period 3; 72 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 1; 8 hours;Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 8 hours;Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Protein; Period 1; 8 hours; 1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 8 hours; 1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Protein; Period 1; 8 hours; 2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 8 hours; 2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Protein; Period 1; 24 hours; Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 24 hours; Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Protein; Period 1; 24 hours; 1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 24 hours; 1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Protein; Period 1; 24 hours;2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 24 hours;2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Protein; Period 1; 48 hours; Trace;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 48 hours; Trace;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Protein; Period 1; 48 hours; 1+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 48 hours; 1+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Protein; Period 1; 48 hours; 2+;n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 48 hours; 2+;n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Protein; Period 1; 72 hours; Trace;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 72 hours; Trace;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Protein; Period 1; 72 hours; 1+;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 72 hours; 1+;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Protein; Period 1; 72 hours; 2+;n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Protein; Period 1; 72 hours; 2+;n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Protein; Period 2; 8 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 8 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 8 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 8 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 8 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 8 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 24 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 24 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 24 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 24 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 24 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 24 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 48 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 48 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 48 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 48 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 48 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 48 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 72 hours; Trace;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 72 hours; Trace;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 72 hours; 1+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 72 hours; 1+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 2; 72 hours; 2+;n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Protein; Period 2; 72 hours; 2+;n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Protein; Period 3; 8 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 8 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 8 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 8 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 8 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 8 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 24 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 24 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 24 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 24 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 24 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 24 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 48 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 48 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 48 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 48 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 48 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 48 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 72 hours; Trace;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 72 hours; Trace;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 72 hours; 1+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 72 hours; 1+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Protein; Period 3; 72 hours; 2+;n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Protein; Period 3; 72 hours; 2+;n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0

11. Primary Outcome: Number of Participants With Urinalysis Dipstick Results for Potential of Hydrogen (pH)-Part A
Description: Urine samples were taken for the assessment of urine pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acid pH (5.0 to 6.0). Dipstick test results for pH were presented as number of participants having pH value as 5, 6, 7, 8 or 9.
Time Frame: 8 hours, 24 hours, 48 hours and 72 hours in Periods 1, 2 and 3
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3439171A 5 mg | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 17 | 6 | 6 | 5 | 6 | 6 | 6
Participants
  Period 1; 8 hours; pH=5; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 8 hours; pH=5; n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Period 1; 8 hours; pH=6; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 8 hours; pH=6; n=6,6,0,0,6,0,0 | 1 | 1 |  |  | 3 |  |
  Period 1; 8 hours; pH=7; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 8 hours; pH=7; n=6,6,0,0,6,0,0 | 3 | 5 |  |  | 2 |  |
  Period 1; 8 hours; pH=8; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 8 hours; pH=8; n=6,6,0,0,6,0,0 | 2 | 0 |  |  | 1 |  |
  Period 1; 8 hours; pH=9; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 8 hours; pH=9; n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Period 1; 24 hours; pH=5; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 24 hours; pH=5; n=6,6,0,0,6,0,0 | 4 | 3 |  |  | 1 |  |
  Period 1; 24 hours; pH=6; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 24 hours; pH=6; n=6,6,0,0,6,0,0 | 2 | 3 |  |  | 3 |  |
  Period 1; 24 hours; pH=7; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 24 hours; pH=7; n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 2 |  |
  Period 1; 24 hours; pH=8; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 24 hours; pH=8; n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Period 1; 24 hours; pH=9; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 24 hours; pH=9; n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Period 1; 48 hours; pH=5; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 48 hours; pH=5; n=6,6,0,0,6,0,0 | 1 | 1 |  |  | 4 |  |
  Period 1; 48 hours; pH=6; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 48 hours; pH=6; n=6,6,0,0,6,0,0 | 4 | 3 |  |  | 2 |  |
  Period 1; 48 hours; pH=7; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 48 hours; pH=7; n=6,6,0,0,6,0,0 | 1 | 2 |  |  | 0 |  |
  Period 1; 48 hours; pH=8; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 48 hours; pH=8; n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Period 1; 48 hours; pH=9; n=6,6,0,0,6,0,0: number analyzed (Participants) | 6 | 6 | 0 | 0 | 6 | 0 | 0
  Period 1; 48 hours; pH=9; n=6,6,0,0,6,0,0 | 0 | 0 |  |  | 0 |  |
  Period 1; 72 hours; pH=5; n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Period 1; 72 hours; pH=5; n=3,0,0,0,6,0,0 | 2 |  |  |  | 2 |  |
  Period 1; 72 hours; pH=6; n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Period 1; 72 hours; pH=6; n=3,0,0,0,6,0,0 | 0 |  |  |  | 4 |  |
  Period 1; 72 hours; pH=7; n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Period 1; 72 hours; pH=7; n=3,0,0,0,6,0,0 | 1 |  |  |  | 0 |  |
  Period 1; 72 hours; pH=8; n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Period 1; 72 hours; pH=8; n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Period 1; 72 hours; pH=9; n=3,0,0,0,6,0,0: number analyzed (Participants) | 3 | 0 | 0 | 0 | 6 | 0 | 0
  Period 1; 72 hours; pH=9; n=3,0,0,0,6,0,0 | 0 |  |  |  | 0 |  |
  Period 2; 8 hours; pH=5; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 8 hours; pH=5; n=6,0,6,0,0,6,0 | 1 |  | 0 |  |  | 0 |
  Period 2; 8 hours; pH=6; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 8 hours; pH=6; n=6,0,6,0,0,6,0 | 2 |  | 0 |  |  | 2 |
  Period 2; 8 hours; pH=7; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 8 hours; pH=7; n=6,0,6,0,0,6,0 | 3 |  | 6 |  |  | 2 |
  Period 2; 8 hours; pH=8; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 8 hours; pH=8; n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 2 |
  Period 2; 8 hours; pH=9; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 8 hours; pH=9; n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Period 2; 24 hours; pH=5; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 24 hours; pH=5; n=6,0,6,0,0,6,0 | 3 |  | 2 |  |  | 3 |
  Period 2; 24 hours; pH=6; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 24 hours; pH=6; n=6,0,6,0,0,6,0 | 3 |  | 3 |  |  | 3 |
  Period 2; 24 hours; pH=7; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 24 hours; pH=7; n=6,0,6,0,0,6,0 | 0 |  | 1 |  |  | 0 |
  Period 2; 24 hours; pH=8; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 24 hours; pH=8; n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Period 2; 24 hours; pH=9; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 24 hours; pH=9; n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  -Period 2; 48 hours; pH=5; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  -Period 2; 48 hours; pH=5; n=6,0,6,0,0,6,0 | 3 |  | 2 |  |  | 4 |
  Period 2; 48 hours; pH=6; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 48 hours; pH=6; n=6,0,6,0,0,6,0 | 2 |  | 1 |  |  | 2 |
  Period 2; 48 hours; pH=7; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 48 hours; pH=7; n=6,0,6,0,0,6,0 | 1 |  | 2 |  |  | 0 |
  Period 2; 48 hours; pH=8; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 48 hours; pH=8; n=6,0,6,0,0,6,0 | 0 |  | 1 |  |  | 0 |
  Period 2; 48 hours; pH=9; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 48 hours; pH=9; n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Period 2; 72 hours; pH=5; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 72 hours; pH=5; n=6,0,6,0,0,6,0 | 1 |  | 1 |  |  | 4 |
  Period 2; 72 hours; pH=6; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 72 hours; pH=6; n=6,0,6,0,0,6,0 | 5 |  | 3 |  |  | 2 |
  Period 2; 72 hours; pH=7; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 72 hours; pH=7; n=6,0,6,0,0,6,0 | 0 |  | 2 |  |  | 0 |
  Period 2; 72 hours; pH=8; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 72 hours; pH=8; n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Period 2; 72 hours; pH=9; n=6,0,6,0,0,6,0: number analyzed (Participants) | 6 | 0 | 6 | 0 | 0 | 6 | 0
  Period 2; 72 hours; pH=9; n=6,0,6,0,0,6,0 | 0 |  | 0 |  |  | 0 |
  Period 3; 8 hours; pH=5; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 8 hours; pH=5; n=5,0,0,5,0,0,6 | 0 |  |  | 1 |  |  | 0
  Period 3; 8 hours; pH=6; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 8 hours; pH=6; n=5,0,0,5,0,0,6 | 1 |  |  | 1 |  |  | 3
  Period 3; 8 hours; pH=7; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 8 hours; pH=7; n=5,0,0,5,0,0,6 | 2 |  |  | 3 |  |  | 1
  Period 3; 8 hours; pH=8; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 8 hours; pH=8; n=5,0,0,5,0,0,6 | 2 |  |  | 0 |  |  | 2
  Period 3; 8 hours; pH=9; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 8 hours; pH=9; n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Period 3; 24 hours; pH=5; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 24 hours; pH=5; n=5,0,0,5,0,0,6 | 2 |  |  | 2 |  |  | 3
  Period 3; 24 hours; pH=6; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 24 hours; pH=6; n=5,0,0,5,0,0,6 | 3 |  |  | 2 |  |  | 3
  Period 3; 24 hours; pH=7; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 24 hours; pH=7; n=5,0,0,5,0,0,6 | 0 |  |  | 1 |  |  | 0
  Period 3; 24 hours; pH=8; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 24 hours; pH=8; n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Period 3; 24 hours; pH=9; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 24 hours; pH=9; n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Period 3; 48 hours; pH=5; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 48 hours; pH=5; n=5,0,0,5,0,0,6 | 2 |  |  | 2 |  |  | 2
  Period 3; 48 hours; pH=6; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 48 hours; pH=6; n=5,0,0,5,0,0,6 | 2 |  |  | 2 |  |  | 4
  Period 3; 48 hours; pH=7; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 48 hours; pH=7; n=5,0,0,5,0,0,6 | 1 |  |  | 1 |  |  | 0
  Period 3; 48 hours; pH=8; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 48 hours; pH=8; n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Period 3; 48 hours; pH=9; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 48 hours; pH=9; n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Period 3; 72 hours; pH=5; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 72 hours; pH=5; n=5,0,0,5,0,0,6 | 1 |  |  | 2 |  |  | 3
  Period 3; 72 hours; pH=6; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 72 hours; pH=6; n=5,0,0,5,0,0,6 | 4 |  |  | 3 |  |  | 3
  Period 3; 72 hours; pH=7; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 72 hours; pH=7; n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Period 3; 72 hours; pH=8; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 72 hours; pH=8; n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0
  Period 3; 72 hours; pH=9; n=5,0,0,5,0,0,6: number analyzed (Participants) | 5 | 0 | 0 | 5 | 0 | 0 | 6
  Period 3; 72 hours; pH=9; n=5,0,0,5,0,0,6 | 0 |  |  | 0 |  |  | 0

12. Primary Outcome: Number of Participants With Abnormal Urinalysis Dipstick Results-Part B
Description: Urine samples were taken for the assessment of following urine parameters: glucose, ketones, OB and protein by dipstick method. The dipstick test gives results in a semi-quantitative manner, and results can be read as Trace, 1+, 2+ indicating proportional concentrations in the urine sample.
Time Frame: Day 2 (24 hours); Day 3 (48 hours); Days 4, 13 and 20 (72 hours); pre-dose on Days 7, 10, 11 and 17
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Glucose; Day2, 24 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day2, 24 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day2, 24 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day3, 48 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day3, 48 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day3, 48 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day4, 72 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day4, 72 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day4, 72 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day7, pre-dose; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day7, pre-dose; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day7, pre-dose; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Glucose; Day10, pre-dose; Trace; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Glucose; Day10, pre-dose; Trace; n=3,0,0,9 | 0 |  |  | 0
  Glucose; Day10, pre-dose; 1+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Glucose; Day10, pre-dose; 1+; n=3,0,0,9 | 0 |  |  | 0
  Glucose; Day10, pre-dose; 2+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Glucose; Day10, pre-dose; 2+; n=3,0,0,9 | 0 |  |  | 0
  Glucose; Day 11, pre-dose; Trace; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Glucose; Day 11, pre-dose; Trace; n=6,9,9,0 | 0 | 0 | 0 |
  Glucose; Day 11, pre-dose; 1+; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Glucose; Day 11, pre-dose; 1+; n=6,9,9,0 | 0 | 0 | 0 |
  Glucose; Day11, pre-dose; 2+; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Glucose; Day11, pre-dose; 2+; n=6,9,9,0 | 0 | 0 | 0 |
  Glucose; Day13, 72 hours; Trace; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Glucose; Day13, 72 hours; Trace; n=3,0,0,9 | 0 |  |  | 0
  Glucose; Day13, 72 hours; 1+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Glucose; Day13, 72 hours; 1+; n=3,0,0,9 | 0 |  |  | 0
  Glucose; Day13, 72 hours; 2+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Glucose; Day13, 72 hours; 2+; n=3,0,0,9 | 0 |  |  | 0
  Glucose; Day17, pre-dose; Trace; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Glucose; Day17, pre-dose; Trace; n=6,9,8,0 | 0 | 0 | 0 |
  Glucose; Day17, pre-dose; 1+; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Glucose; Day17, pre-dose; 1+; n=6,9,8,0 | 0 | 0 | 0 |
  Glucose; Day17, pre-dose; 2+; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Glucose; Day17, pre-dose; 2+; n=6,9,8,0 | 0 | 0 | 0 |
  Glucose; Day20, 72 hours; Trace; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Glucose; Day20, 72 hours; Trace; n=6,9,7,0 | 0 | 0 | 0 |
  Glucose; Day20, 72 hours; 1+; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Glucose; Day20, 72 hours; 1+; n=6,9,7,0 | 0 | 0 | 0 |
  Glucose; Day20, 72 hours; 2+; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Glucose; Day20, 72 hours; 2+; n=6,9,7,0 | 0 | 0 | 0 |
  Ketones; Day2, 24 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day2, 24 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day2, 24 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day3, 48 hours; Trace; ; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day3, 48 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day3, 48 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day4, 72 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day4, 72 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day4, 72 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day7, pre-dose; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day7, pre-dose; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day7, pre-dose; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Ketones; Day10, pre-dose; Trace; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Ketones; Day10, pre-dose; Trace; n=3,0,0,9 | 0 |  |  | 0
  Ketones; Day10, pre-dose; 1+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Ketones; Day10, pre-dose; 1+; n=3,0,0,9 | 0 |  |  | 0
  Ketones; Day10, pre-dose; 2+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Ketones; Day10, pre-dose; 2+; n=3,0,0,9 | 0 |  |  | 0
  Ketones; Day 11, pre-dose; Trace; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Ketones; Day 11, pre-dose; Trace; n=6,9,9,0 | 0 | 1 | 0 |
  Ketones; Day11, pre-dose; 1+; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Ketones; Day11, pre-dose; 1+; n=6,9,9,0 | 0 | 0 | 0 |
  Ketones; Day11, pre-dose; 2+; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Ketones; Day11, pre-dose; 2+; n=6,9,9,0 | 0 | 0 | 0 |
  Ketones; Day13, 72 hours; Trace; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Ketones; Day13, 72 hours; Trace; n=3,0,0,9 | 0 |  |  | 0
  Ketones; Day13, 72 hours; 1+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Ketones; Day13, 72 hours; 1+; n=3,0,0,9 | 0 |  |  | 0
  Ketones; Day13, 72 hours; 2+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Ketones; Day13, 72 hours; 2+; n=3,0,0,9 | 0 |  |  | 0
  Ketones; Day17, pre-dose; Trace; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Ketones; Day17, pre-dose; Trace; n=6,9,8,0 | 0 | 0 | 0 |
  Ketones; Day17, pre-dose; 1+; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Ketones; Day17, pre-dose; 1+; n=6,9,8,0 | 0 | 0 | 0 |
  Ketones; Day17, pre-dose; 2+; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Ketones; Day17, pre-dose; 2+; n=6,9,8,0 | 0 | 0 | 0 |
  Ketones; Day20, 72 hours; Trace; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Ketones; Day20, 72 hours; Trace; n=6,9,7,0 | 0 | 0 | 0 |
  Ketones; Day20, 72 hours; 1+; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Ketones; Day20, 72 hours; 1+; n=6,9,7,0 | 0 | 0 | 0 |
  Ketones; Day20, 72 hours; 2+; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Ketones; Day20, 72 hours; 2+; n=6,9,7,0 | 0 | 0 | 0 |
  OB; Day2, 24 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  OB; Day2, 24 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  OB; Day2, 24 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  OB; Day3, 48 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  OB; Day3, 48 hours; 1+; n=9,9,9,9 | 1 | 0 | 0 | 2
  OB; Day3, 48 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  OB; Day4, 72 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  OB; Day4, 72 hours; 1+; n=9,9,9,9 | 0 | 0 | 1 | 0
  OB; Day4, 72 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  OB; Day7, pre-dose; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  OB; Day7, pre-dose; 1+; n=9,9,9,9 | 0 | 0 | 1 | 0
  OB; Day7, pre-dose; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  OB; Day10, pre-dose; Trace; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  OB; Day10, pre-dose; Trace; n=3,0,0,9 | 0 |  |  | 0
  OB; Day10, pre-dose; 1+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  OB; Day10, pre-dose; 1+; n=3,0,0,9 | 0 |  |  | 0
  OB; Day10, pre-dose; 2+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  OB; Day10, pre-dose; 2+; n=3,0,0,9 | 0 |  |  | 0
  OB; Day 11, pre-dose; Trace; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  OB; Day 11, pre-dose; Trace; n=6,9,9,0 | 0 | 0 | 0 |
  OB; Day11, pre-dose; 1+; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  OB; Day11, pre-dose; 1+; n=6,9,9,0 | 0 | 0 | 1 |
  OB; Day11, pre-dose; 2+; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  OB; Day11, pre-dose; 2+; n=6,9,9,0 | 0 | 0 | 0 |
  OB; Day13, 72 hours; Trace; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  OB; Day13, 72 hours; Trace; n=3,0,0,9 | 0 |  |  | 0
  OB; Day13, 72 hours; 1+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  OB; Day13, 72 hours; 1+; n=3,0,0,9 | 0 |  |  | 1
  OB; Day13, 72 hours; 2+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  OB; Day13, 72 hours; 2+; n=3,0,0,9 | 0 |  |  | 0
  OB; Day17, pre-dose; Trace; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  OB; Day17, pre-dose; Trace; n=6,9,8,0 | 0 | 0 | 0 |
  OB; Day17, pre-dose; 1+; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  OB; Day17, pre-dose; 1+; n=6,9,8,0 | 1 | 0 | 1 |
  OB; Day17, pre-dose; 2+; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  OB; Day17, pre-dose; 2+; n=6,9,8,0 | 0 | 0 | 0 |
  OB; Day20, 72 hours; Trace; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  OB; Day20, 72 hours; Trace; n=6,9,7,0 | 0 | 0 | 0 |
  OB; Day20, 72 hours; 1+; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  OB; Day20, 72 hours; 1+; n=6,9,7,0 | 1 | 0 | 2 |
  OB; Day20, 72 hours; 2+; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  OB; Day20, 72 hours; 2+; n=6,9,7,0 | 0 | 0 | 0 |
  Protein; Day2, 24 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day2, 24 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day2, 24 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day3, 48 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day3, 48 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day3, 48 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day4, 72 hours; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day4, 72 hours; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day4, 72 hours; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day7, pre-dose; Trace; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day7, pre-dose; 1+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day7, pre-dose; 2+; n=9,9,9,9 | 0 | 0 | 0 | 0
  Protein; Day10, pre-dose; Trace; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Protein; Day10, pre-dose; Trace; n=3,0,0,9 | 0 |  |  | 0
  Protein; Day10, pre-dose; 1+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Protein; Day10, pre-dose; 1+; n=3,0,0,9 | 0 |  |  | 0
  Protein; Day10, pre-dose; 2+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Protein; Day10, pre-dose; 2+; n=3,0,0,9 | 0 |  |  | 0
  Protein; Day 11, pre-dose; Trace; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Protein; Day 11, pre-dose; Trace; n=6,9,9,0 | 0 | 0 | 0 |
  Protein; Day11, pre-dose; 1+; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Protein; Day11, pre-dose; 1+; n=6,9,9,0 | 0 | 0 | 0 |
  Protein; Day11, pre-dose; 2+; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Protein; Day11, pre-dose; 2+; n=6,9,9,0 | 0 | 0 | 0 |
  Protein; Day13, 72 hours; Trace; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Protein; Day13, 72 hours; Trace; n=3,0,0,9 | 0 |  |  | 0
  Protein; Day13, 72 hours; 1+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Protein; Day13, 72 hours; 1+; n=3,0,0,9 | 0 |  |  | 0
  Protein; Day13, 72 hours; 2+; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Protein; Day13, 72 hours; 2+; n=3,0,0,9 | 0 |  |  | 0
  Protein; Day17, pre-dose; Trace; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Protein; Day17, pre-dose; Trace; n=6,9,8,0 | 0 | 0 | 0 |
  Protein; Day17, pre-dose; 1+; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Protein; Day17, pre-dose; 1+; n=6,9,8,0 | 0 | 0 | 0 |
  Protein; Day17, pre-dose; 2+; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Protein; Day17, pre-dose; 2+; n=6,9,8,0 | 0 | 0 | 0 |
  Protein; Day20, 72 hours; Trace; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Protein; Day20, 72 hours; Trace; n=6,9,7,0 | 0 | 0 | 0 |
  Protein; Day20, 72 hours; 1+; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Protein; Day20, 72 hours; 1+; n=6,9,7,0 | 0 | 0 | 0 |
  Protein; Day20, 72 hours; 2+; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Protein; Day20, 72 hours; 2+; n=6,9,7,0 | 0 | 0 | 0 |

13. Primary Outcome: Number of Participants With Urinalysis Dipstick Results (pH)-Part B
Description: as for outcome 11
Time Frame: Day 2 (24 hours); Day 3 (48 hours); Days 4, 13 and 20 (72 hours); pre-dose on Days 7, 10, 11 and 17
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  Day2, 24 hours; pH=5; n=9,9,9,9 | 1 | 2 | 1 | 1
  Day2, 24 hours; pH=6; n=9,9,9,9 | 4 | 5 | 5 | 8
  Day2, 24 hours; pH=7; n=9,9,9,9 | 4 | 2 | 2 | 0
  Day2, 24 hours; pH=8; n=9,9,9,9 | 0 | 0 | 1 | 0
  Day2, 24 hours; pH=9; n=9,9,9,9 | 0 | 0 | 0 | 0
  Day3, 48 hours; pH=5; n=9,9,9,9 | 1 | 4 | 4 | 3
  Day3, 48 hours; pH=6; n=9,9,9,9 | 6 | 4 | 3 | 6
  Day3, 48 hours; pH=7; n=9,9,9,9 | 2 | 0 | 2 | 0
  Day3, 48 hours; pH=8; n=9,9,9,9 | 0 | 1 | 0 | 0
  Day3, 48 hours; pH=9; n=9,9,9,9 | 0 | 0 | 0 | 0
  Day4, 72 hours; pH=5; n=9,9,9,9 | 1 | 3 | 4 | 3
  Day4, 72 hours; pH=6; n=9,9,9,9 | 5 | 3 | 5 | 5
  Day4, 72 hours; pH=7; n=9,9,9,9 | 3 | 3 | 0 | 1
  Day4, 72 hours; pH=8; n=9,9,9,9 | 0 | 0 | 0 | 0
  Day4, 72 hours; pH=9; n=9,9,9,9 | 0 | 0 | 0 | 0
  Day7, pre-dose; pH=5; n=9,9,9,9 | 1 | 3 | 4 | 2
  Day7, pre-dose; pH=6; n=9,9,9,9 | 3 | 5 | 5 | 5
  Day7, pre-dose; pH=7; n=9,9,9,9 | 5 | 1 | 0 | 1
  Day7, pre-dose; pH=8; n=9,9,9,9 | 0 | 0 | 0 | 1
  Day7, pre-dose; pH=9; n=9,9,9,9 | 0 | 0 | 0 | 0
  Day10, pre-dose; pH=5; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day10, pre-dose; pH=5; n=3,0,0,9 | 1 |  |  | 4
  Day10, pre-dose; pH=6; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day10, pre-dose; pH=6; n=3,0,0,9 | 2 |  |  | 4
  Day10, pre-dose; pH=7; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day10, pre-dose; pH=7; n=3,0,0,9 | 0 | 0 |  | 1
  Day10, pre-dose; pH=8; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day10, pre-dose; pH=8; n=3,0,0,9 | 0 |  |  | 0
  Day10, pre-dose; pH=9; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day10, pre-dose; pH=9; n=3,0,0,9 | 0 |  |  | 0
  Day 11, pre-dose; pH=5; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Day 11, pre-dose; pH=5; n=6,9,9,0 | 0 | 3 | 3 |
  Day 11, pre-dose; pH=6; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Day 11, pre-dose; pH=6; n=6,9,9,0 | 3 | 5 | 4 |
  Day 11, pre-dose; pH=7; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Day 11, pre-dose; pH=7; n=6,9,9,0 | 3 | 1 | 2 |
  Day 11, pre-dose; pH=8; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Day 11, pre-dose; pH=8; n=6,9,9,0 | 0 | 0 | 0 |
  Day 11, pre-dose; pH=9; n=6,9,9,0: number analyzed (Participants) | 6 | 9 | 9 | 0
  Day 11, pre-dose; pH=9; n=6,9,9,0 | 0 | 0 | 0 |
  Day13, 72 hours; pH=5; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day13, 72 hours; pH=5; n=3,0,0,9 | 0 |  |  | 4
  Day13, 72 hours; pH=6; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day13, 72 hours; pH=6; n=3,0,0,9 | 2 |  |  | 2
  Day13, 72 hours; pH=7; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day13, 72 hours; pH=7; n=3,0,0,9 | 1 |  |  | 3
  Day13, 72 hours; pH=8; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day13, 72 hours; pH=8; n=3,0,0,9 | 0 |  |  | 0
  Day13, 72 hours; pH=9; n=3,0,0,9: number analyzed (Participants) | 3 | 0 | 0 | 9
  Day13, 72 hours; pH=9; n=3,0,0,9 | 0 |  |  | 0
  Day17, pre-dose; pH=5; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Day17, pre-dose; pH=5; n=6,9,8,0 | 1 | 1 | 3 |
  Day17, pre-dose; pH=6; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Day17, pre-dose; pH=6; n=6,9,8,0 | 1 | 6 | 3 |
  Day17, pre-dose; pH=7; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Day17, pre-dose; pH=7; n=6,9,8,0 | 4 | 2 | 2 |
  Day17, pre-dose; pH=8; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Day17, pre-dose; pH=8; n=6,9,8,0 | 0 | 0 | 0 |
  Day17, pre-dose; pH=9; n=6,9,8,0: number analyzed (Participants) | 6 | 9 | 8 | 0
  Day17, pre-dose; pH=9; n=6,9,8,0 | 0 | 0 | 0 |
  Day20, 72 hours; pH=5; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Day20, 72 hours; pH=5; n=6,9,7,0 | 1 | 2 | 4 |
  Day20, 72 hours; pH=6; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Day20, 72 hours; pH=6; n=6,9,7,0 | 2 | 5 | 3 |
  Day20, 72 hours; pH=7; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Day20, 72 hours; pH=7; n=6,9,7,0 | 3 | 2 | 0 |
  Day20, 72 hours; pH=8; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Day20, 72 hours; pH=8; n=6,9,7,0 | 0 | 0 | 0 |
  Day20, 72 hours; pH=9; n=6,9,7,0: number analyzed (Participants) | 6 | 9 | 7 | 0
  Day20, 72 hours; pH=9; n=6,9,7,0 | 0 | 0 | 0 |

14. Primary Outcome: Number of Participants With Abnormal Urinalysis Dipstick Results-Part C
Description: as for outcome 12
Time Frame: 8 hours, 24 hours, 48 hours and 72 hours in Period 1 and Period 2
Population: Safety Population. All participants in Part C (11, 11) were included in the analysis; however, only participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Participants
  Glucose; Period 1, 8 hours; Trace; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 8 hours; Trace; n=6, 6 | 0 | 0
  Glucose; Period 1, 8 hours; 1+; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 8 hours; 1+; n=6, 6 | 0 | 0
  Glucose; Period 1, 8 hours; 2+; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 8 hours; 2+; n=6, 6 | 0 | 0
  Glucose; Period 1, 24 hours; Trace; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 24 hours; Trace; n=6, 6 | 0 | 0
  Glucose; Period 1, 24 hours; 1+; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 24 hours; 1+; n=6, 6 | 0 | 0
  Glucose; Period 1, 24 hours; 2+; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 24 hours; 2+; n=6, 6 | 0 | 0
  Glucose; Period 1, 48 hours; Trace; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 48 hours; Trace; n=6, 6 | 0 | 0
  Glucose; Period 1, 48 hours; 1+; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 48 hours; 1+; n=6, 6 | 0 | 0
  Glucose; Period 1, 48 hours; 2+; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 48 hours; 2+; n=6, 6 | 0 | 0
  Glucose; Period 1, 72 hours; Trace; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 72 hours; Trace; n=6, 6 | 0 | 0
  Glucose; Period 1, 72 hours; 1+; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 72 hours; 1+; n=6, 6 | 0 | 0
  Glucose; Period 1, 72 hours; 2+; n=6, 6: number analyzed (Participants) | 6 | 6
  Glucose; Period 1, 72 hours; 2+; n=6, 6 | 0 | 0
  Glucose; Period 2, 8 hours; Trace; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 8 hours; Trace; n=5, 5 | 0 | 0
  Glucose; Period 2, 8 hours; 1+; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 8 hours; 1+; n=5, 5 | 0 | 0
  Glucose; Period 2, 8 hours; 2+;n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 8 hours; 2+;n=5, 5 | 0 | 0
  Glucose; Period 2, 24 hours; Trace; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 24 hours; Trace; n=5, 5 | 0 | 0
  Glucose; Period 2, 24 hours; 1+; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 24 hours; 1+; n=5, 5 | 0 | 0
  Glucose; Period 2, 24 hours; 2+; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 24 hours; 2+; n=5, 5 | 0 | 0
  Glucose; Period 2, 48 hours; Trace; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 48 hours; Trace; n=5, 5 | 0 | 0
  Glucose; Period 2, 48 hours; 1+; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 48 hours; 1+; n=5, 5 | 0 | 0
  Glucose; Period 2, 48 hours; 2+; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 48 hours; 2+; n=5, 5 | 0 | 0
  Glucose; Period 2, 72 hours; Trace; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 72 hours; Trace; n=5, 5 | 0 | 0
  Glucose; Period 2, 72 hours; 1+; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 72 hours; 1+; n=5, 5 | 0 | 0
  Glucose; Period 2, 72 hours; 2+; n=5, 5: number analyzed (Participants) | 5 | 5
  Glucose; Period 2, 72 hours; 2+; n=5, 5 | 0 | 0
  Ketone; Period 1, 8 hours; Trace; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 8 hours; Trace; n=6,6 | 0 | 0
  Ketone; Period 1, 8 hours; 1+; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 8 hours; 1+; n=6,6 | 0 | 0
  Ketone; Period 1, 8 hours; 2+; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 8 hours; 2+; n=6,6 | 0 | 0
  Ketone; Period 1, 24 hours; Trace; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 24 hours; Trace; n=6,6 | 0 | 0
  Ketone; Period 1, 24 hours; 1+; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 24 hours; 1+; n=6,6 | 0 | 0
  Ketone; Period 1, 24 hours; 2+; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 24 hours; 2+; n=6,6 | 0 | 0
  Ketone; Period 1, 48 hours; Trace; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 48 hours; Trace; n=6,6 | 1 | 0
  Ketone; Period 1, 48 hours; 1+; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 48 hours; 1+; n=6,6 | 0 | 0
  Ketone; Period 1, 48 hours; 2+; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 48 hours; 2+; n=6,6 | 0 | 0
  Ketone; Period 1, 72 hours; Trace; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 72 hours; Trace; n=6,6 | 0 | 0
  Ketone; Period 1, 72 hours; 1+; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 72 hours; 1+; n=6,6 | 0 | 1
  Ketone; Period 1, 72 hours; 2+; n=6,6: number analyzed (Participants) | 6 | 6
  Ketone; Period 1, 72 hours; 2+; n=6,6 | 0 | 0
  Ketone; Period 2, 8 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 8 hours; Trace; n=5,5 | 0 | 0
  Ketone; Period 2, 8 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 8 hours; 1+; n=5,5 | 0 | 0
  Ketone; Period 2, 8 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 8 hours; 2+; n=5,5 | 0 | 0
  Ketone; Period 2, 24 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 24 hours; Trace; n=5,5 | 0 | 0
  Ketone; Period 2, 24 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 24 hours; 1+; n=5,5 | 0 | 0
  Ketone; Period 2, 24 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 24 hours; 2+; n=5,5 | 0 | 0
  Ketone; Period 2, 48 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 48 hours; Trace; n=5,5 | 0 | 1
  Ketone; Period 2, 48 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 48 hours; 1+; n=5,5 | 0 | 0
  Ketone; Period 2, 48 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 48 hours; 2+; n=5,5 | 0 | 0
  Ketone; Period 2, 72 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 72 hours; Trace; n=5,5 | 0 | 1
  Ketone; Period 2, 72 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 72 hours; 1+; n=5,5 | 0 | 0
  Ketone; Period 2, 72 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  Ketone; Period 2, 72 hours; 2+; n=5,5 | 0 | 0
  OB; Period 1, 8 hours; Trace; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 8 hours; Trace; n=6, 6 | 0 | 0
  OB; Period 1, 8 hours; 1+; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 8 hours; 1+; n=6, 6 | 1 | 0
  OB; Period 1, 8 hours; 2+; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 8 hours; 2+; n=6, 6 | 0 | 0
  OB; Period 1, 24 hours; Trace; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 24 hours; Trace; n=6, 6 | 0 | 0
  OB; Period 1, 24 hours; 1+; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 24 hours; 1+; n=6, 6 | 1 | 0
  OB; Period 1, 24 hours; 2+; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 24 hours; 2+; n=6, 6 | 0 | 0
  OB; Period 1, 48 hours; Trace; n=6,6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 48 hours; Trace; n=6,6 | 0 | 0
  OB; Period 1, 48 hours; 1+; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 48 hours; 1+; n=6, 6 | 1 | 0
  OB; Period 1, 48 hours; 2+; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 48 hours; 2+; n=6, 6 | 0 | 0
  OB; Period 1, 72 hours; Trace; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 72 hours; Trace; n=6, 6 | 0 | 0
  OB; Period 1, 72 hours; 1+; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 72 hours; 1+; n=6, 6 | 2 | 1
  OB; Period 1, 72 hours; 2+; n=6, 6: number analyzed (Participants) | 6 | 6
  OB; Period 1, 72 hours; 2+; n=6, 6 | 0 | 0
  OB; Period 2, 8 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 8 hours; Trace; n=5,5 | 0 | 0
  OB; Period 2, 8 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 8 hours; 1+; n=5,5 | 0 | 0
  OB; Period 2, 8 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 8 hours; 2+; n=5,5 | 0 | 1
  OB; Period 2, 24 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 24 hours; Trace; n=5,5 | 0 | 0
  OB; Period 2, 24 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 24 hours; 1+; n=5,5 | 1 | 1
  OB; Period 2, 24 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 24 hours; 2+; n=5,5 | 0 | 0
  OB; Period 2, 48 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 48 hours; Trace; n=5,5 | 0 | 0
  OB; Period 2, 48 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 48 hours; 1+; n=5,5 | 1 | 1
  OB; Period 2, 48 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 48 hours; 2+; n=5,5 | 0 | 0
  OB; Period 2, 72 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 72 hours; Trace; n=5,5 | 0 | 0
  OB; Period 2, 72 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 72 hours; 1+; n=5,5 | 1 | 1
  OB; Period 2, 72 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  OB; Period 2, 72 hours; 2+; n=5,5 | 0 | 0
  Protein; Period 1, 8 hours; Trace; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 8 hours; Trace; n=6,6 | 0 | 0
  Protein; Period 1, 8 hours; 1+; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 8 hours; 1+; n=6,6 | 0 | 0
  Protein; Period 1, 8 hours; 2+; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 8 hours; 2+; n=6,6 | 0 | 0
  Protein; Period 1, 24 hours; Trace; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 24 hours; Trace; n=6,6 | 0 | 0
  Protein; Period 1, 24 hours; 1+; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 24 hours; 1+; n=6,6 | 0 | 0
  Protein; Period 1, 24 hours; 2+; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 24 hours; 2+; n=6,6 | 0 | 0
  Protein; Period 1, 48 hours; Trace; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 48 hours; Trace; n=6,6 | 0 | 0
  Protein; Period 1, 48 hours; 1+; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 48 hours; 1+; n=6,6 | 0 | 0
  Protein; Period 1, 48 hours; 2+; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 48 hours; 2+; n=6,6 | 0 | 0
  Protein; Period 1, 72 hours; Trace; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 72 hours; Trace; n=6,6 | 0 | 0
  Protein; Period 1, 72 hours; 1+; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 72 hours; 1+; n=6,6 | 0 | 0
  Protein; Period 1, 72 hours; 2+; n=6,6: number analyzed (Participants) | 6 | 6
  Protein; Period 1, 72 hours; 2+; n=6,6 | 0 | 0
  Protein; Period 2, 8 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 8 hours; Trace; n=5,5 | 0 | 0
  Protein; Period 2, 8 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 8 hours; 1+; n=5,5 | 0 | 0
  Protein; Period 2, 8 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 8 hours; 2+; n=5,5 | 0 | 0
  Protein; Period 2, 24 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 24 hours; Trace; n=5,5 | 0 | 0
  Protein; Period 2, 24 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 24 hours; 1+; n=5,5 | 0 | 0
  Protein; Period 2, 24 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 24 hours; 2+; n=5,5 | 0 | 0
  Protein; Period 2, 48 hours; Trace;n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 48 hours; Trace;n=5,5 | 0 | 0
  Protein; Period 2, 48 hours; 1+;n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 48 hours; 1+;n=5,5 | 0 | 0
  Protein; Period 2, 48 hours; 2+;n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 48 hours; 2+;n=5,5 | 0 | 0
  Protein; Period 2, 72 hours; Trace; n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 72 hours; Trace; n=5,5 | 0 | 0
  Protein; Period 2, 72 hours; 1+; n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 72 hours; 1+; n=5,5 | 0 | 0
  Protein; Period 2, 72 hours; 2+; n=5,5: number analyzed (Participants) | 5 | 5
  Protein; Period 2, 72 hours; 2+; n=5,5 | 0 | 0

15. Primary Outcome: Number of Participants With Urinalysis Dipstick Results (pH)-Part C
Description: as for outcome 11
Time Frame: 8 hours, 24 hours, 48 hours and 72 hours in Period 1 and Period 2
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Participants
  Period 1, 8 hours; pH=5; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 8 hours; pH=5; n=6,6 | 0 | 1
  Period 1, 8 hours; pH=6; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 8 hours; pH=6; n=6,6 | 1 | 1
  Period 1, 8 hours; pH=7; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 8 hours; pH=7; n=6,6 | 3 | 4
  Period 1, 8 hours; pH=8; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 8 hours; pH=8; n=6,6 | 2 | 0
  Period 1, 8 hours; pH=9; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 8 hours; pH=9; n=6,6 | 0 | 0
  Period 1, 24 hours; pH=5; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 24 hours; pH=5; n=6,6 | 2 | 2
  Period 1, 24 hours; pH=6; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 24 hours; pH=6; n=6,6 | 3 | 4
  Period 1, 24 hours; pH=7; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 24 hours; pH=7; n=6,6 | 1 | 0
  Period 1, 24 hours; pH=8; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 24 hours; pH=8; n=6,6 | 0 | 0
  Period 1, 24 hours; pH=9; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 24 hours; pH=9; n=6,6 | 0 | 0
  Period 1, 48 hours; pH=5; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 48 hours; pH=5; n=6,6 | 2 | 4
  Period 1, 48 hours; pH=6; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 48 hours; pH=6; n=6,6 | 3 | 2
  Period 1, 48 hours; pH=7; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 48 hours; pH=7; n=6,6 | 1 | 0
  Period 1, 48 hours; pH=8; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 48 hours; pH=8; n=6,6 | 0 | 0
  Period 1, 48 hours; pH=9; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 48 hours; pH=9; n=6,6 | 0 | 0
  Period 1, 72 hours; pH=5; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 72 hours; pH=5; n=6,6 | 3 | 3
  Period 1, 72 hours; pH=6; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 72 hours; pH=6; n=6,6 | 3 | 3
  Period 1, 72 hours; pH=7; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 72 hours; pH=7; n=6,6 | 0 | 0
  Period 1, 72 hours; pH=8; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 72 hours; pH=8; n=6,6 | 0 | 0
  Period 1, 72 hours; pH=9; n=6,6: number analyzed (Participants) | 6 | 6
  Period 1, 72 hours; pH=9; n=6,6 | 0 | 0
  Period 2, 8 hours; pH=5; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 8 hours; pH=5; n=5,5 | 1 | 1
  Period 2, 8 hours; pH=6; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 8 hours; pH=6; n=5,5 | 1 | 1
  Period 2, 8 hours; pH=7; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 8 hours; pH=7; n=5,5 | 3 | 3
  Period 2, 8 hours; pH=8; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 8 hours; pH=8; n=5,5 | 0 | 0
  Period 2, 8 hours; pH=9; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 8 hours; pH=9; n=5,5 | 0 | 0
  Period 2, 24 hours; pH=5; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 24 hours; pH=5; n=5,5 | 3 | 0
  Period 2, 24 hours; pH=6; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 24 hours; pH=6; n=5,5 | 1 | 5
  Period 2, 24 hours; pH=7; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 24 hours; pH=7; n=5,5 | 1 | 0
  Period 2, 24 hours; pH=8; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 24 hours; pH=8; n=5,5 | 0 | 0
  Period 2, 24 hours; pH=9; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 24 hours; pH=9; n=5,5 | 0 | 0
  Period 2, 48 hours; pH=5; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 48 hours; pH=5; n=5,5 | 3 | 0
  Period 2, 48 hours; pH=6; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 48 hours; pH=6; n=5,5 | 2 | 4
  Period 2, 48 hours; pH=7; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 48 hours; pH=7; n=5,5 | 0 | 1
  Period 2, 48 hours; pH=8; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 48 hours; pH=8; n=5,5 | 0 | 0
  Period 2, 48 hours; pH=9; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 48 hours; pH=9; n=5,5 | 0 | 0
  Period 2, 72 hours; pH=5; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 72 hours; pH=5; n=5,5 | 2 | 1
  Period 2, 72 hours; pH=6; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 72 hours; pH=6; n=5,5 | 3 | 4
  Period 2, 72 hours; pH=7; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 72 hours; pH=7; n=5,5 | 0 | 0
  Period 2, 72 hours; pH=8; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 72 hours; pH=8; n=5,5 | 0 | 0
  Period 2, 72 hours; pH=9; n=5,5: number analyzed (Participants) | 5 | 5
  Period 2, 72 hours; pH=9; n=5,5 | 0 | 0

16. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance-Part A
Description: Vital signs were measured in a supine position after five minutes of rest and included temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate and respiratory rate. The clinical concern range for the parameters included: SBP (low: <85 millimeters of mercury [mmHg] and high: >160 mmHg), DBP (low: <45 mmHg and high: >100 mmHg) and heart rate (low: <40 beats per minute [bpm] and high: >110 bpm). Number of participants with any vital signs of potential clinical importance is reported.
Time Frame: Up to Day 40
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3439171A 5 mg | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 17 | 6 | 6 | 5 | 6 | 6 | 6
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 1

17. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance-Part B
Description: Vital signs were measured in a supine position after five minutes of rest and included temperature, SBP, DBP, heart rate and respiratory rate. The clinical concern range for the parameters included: SBP (low: <85 mmHg and high: >160 mmHg), DBP (low: <45 mmHg and high: >100 mmHg) and heart rate (low: <40 bpm and high: >110 bpm). Number of participants with any vital signs of potential clinical importance is reported.
Time Frame: Up to Day 34
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants | 0 | 0 | 0 | 2

18. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance-Part C
Description: as for outcome 17
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Participants | 1 | 0

19. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings-Part A
Description: Twelve-lead ECGs were recorded with the participants in a supine position using an ECG machine that automatically calculated heart rate and measured PR, QRS, QT and corrected QT (QTc) intervals. Clinically significant (CS) and not clinically significant (NCS) abnormal ECG findings have been presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for worst case post-Baseline is presented. Baseline value is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Up to Day 40
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: GSK3439171A 5 mg | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 17 | 6 | 6 | 5 | 6 | 6 | 6
Participants
  NCS | 16 | 5 | 6 | 5 | 4 | 6 | 6
  CS | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Primary Outcome: Number of Participants With Abnormal ECG Findings-Part B
Description: Twelve-lead ECGs were recorded with the participants in a supine position using an ECG machine that automatically calculated heart rate and measured PR, QRS, QT and QTc intervals. CS and NCS abnormal ECG findings have been presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for worst case post-Baseline is presented. Baseline value is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Up to Day 34
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Placebo | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9 | 9 | 9 | 9
Participants
  NCS | 9 | 9 | 8 | 9
  CS | 0 | 0 | 0 | 0

21. Primary Outcome: Number of Participants With Abnormal ECG Findings-Part C
Description: as for outcome 20
Time Frame: Up to Day 29
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Participants
  NCS | 10 | 11
  CS | 0 | 0

22. Primary Outcome: Area Under Tha Plasma Drug Concentration Versus Time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC[0 to t]) of GSK3439171A Following Single Dose-Part A (GSK3439171A 5 mg Only)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis.
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36 and 48 hours post-dose
Population: Pharmacokinetic Population comprised of participants in the Safety population for whom a Pharmacokinetic sample was taken and analyzed for GSK3439171A and result reported
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part A: GSK3439171A 5 mg
Number analyzed (Participants) | 6
Hours*nanograms per milliliter | 1180.6 (48.9)

23. Primary Outcome: AUC(0 to t) of GSK3439171A Following Single Dose-Part A (GSK3439171A 10 mg, 30 mg, 60 mg, 120 mg and 180 mg)
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
Hours*nanograms per milliliter | 2268.6 (34.4) | 9289.4 (22.3) | 17052.3 (27.9) | 35822.0 (25.3) | 46086.3 (14.4)

24. Primary Outcome: AUC(0 to t) of GSK3439171A Following Single Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 9
Hours*nanograms per milliliter | 1474.0 (24.6) | 2299.2 (31.5)

25. Primary Outcome: AUC(0 to t) of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 7
Hours*nanograms per milliliter | 2072.8 (30.7) | 3628.1 (39.6)

26. Primary Outcome: AUC(0 to t) of GSK3439171A Following Single Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Hours*nanograms per milliliter | 10031.8 (24.5)

27. Primary Outcome: AUC(0 to t) of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 10 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Hours*nanograms per milliliter | 14896.5 (26.4)

28. Primary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC[0 to Inf]) of GSK3439171A Following Single Dose-Part A (GSK3439171A 5 mg Only)
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36 and 48 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part A: GSK3439171A 5 mg
Number analyzed (Participants) | 6
Hours*nanograms per milliliter | 1247.2 (51.9)

29. Primary Outcome: AUC(0 to Inf) of GSK3439171A Following Single Dose-Part A (GSK3439171A 10 mg, 30 mg, 60 mg, 120 mg and 180 mg)
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
Hours*nanograms per milliliter | 2305.3 (34.5) | 9441.8 (22.2) | 17257.9 (28.7) | 36478.0 (26.1) | 46844.6 (15.2)

30. Primary Outcome: AUC(0 to Inf) of GSK3439171A Following Single Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 9
Hours*nanograms per milliliter | 1514.9 (25.1) | 2345.6 (31.7)

31. Primary Outcome: AUC(0 to Inf) of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 7
Hours*nanograms per milliliter | 2129.0 (31.8) | 3687.1 (40.2)

32. Primary Outcome: AUC(0 to Inf) of GSK3439171A Following Single Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Hours*nanograms per milliliter | 10182.6 (24.9)

33. Primary Outcome: AUC(0 to Inf) of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 10 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Hours*nanograms per milliliter | 15098.7 (27.3)

34. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK3439171A Following Single Dose-Part A (GSK3439171A 5 mg Only)
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36 and 48 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part A: GSK3439171A 5 mg
Number analyzed (Participants) | 6
Nanograms per milliliter | 111.01 (10.9)

35. Primary Outcome: Cmax of GSK3439171A Following Single Dose-Part A (GSK3439171A 10 mg, 30 mg, 60 mg, 120 mg and 180 mg)
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
Nanograms per milliliter | 214.03 (28.1) | 635.37 (26.8) | 1272.26 (19.4) | 2132.49 (19.1) | 2938.01 (21.2)

36. Primary Outcome: Cmax of GSK3439171A Following Single Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 9
Nanograms per milliliter | 117.40 (25.1) | 192.62 (20.8)

37. Primary Outcome: Cmax of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 7
Nanograms per milliliter | 138.08 (19.3) | 243.98 (28.0)

38. Primary Outcome: Cmax of GSK3439171A Following Single Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Nanograms per milliliter | 682.62 (24.8)

39. Primary Outcome: Cmax of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 10 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Nanograms per milliliter | 1016.29 (24.3)

40. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of GSK3439171A Following Single Dose-Part A (GSK3439171A 5 mg Only)
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36 and 48 hours post-dose
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: GSK3439171A 5 mg
Number analyzed (Participants) | 6
Hours | 1.0000 [0.500 to 6.000]

41. Primary Outcome: Tmax of GSK3439171A Following Single Dose-Part A (GSK3439171A 10 mg, 30 mg, 60 mg, 120 mg and 180 mg)
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
Hours | 0.9830 [0.500 to 4.000] | 1.5000 [0.500 to 3.000] | 1.7415 [0.500 to 3.000] | 4.0000 [2.017 to 4.000] | 2.9915 [1.650 to 4.000]

42. Primary Outcome: Tmax of GSK3439171A Following Single Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 9
Hours | 1.5000 [0.483 to 4.000] | 2.0000 [1.500 to 3.983]

43. Primary Outcome: Tmax of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 7
Hours | 3.0000 [1.000 to 4.000] | 2.0000 [2.000 to 4.000]

44. Primary Outcome: Tmax of GSK3439171A Following Single Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Hours | 4.0000 [1.483 to 6.000]

45. Primary Outcome: Tmax of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 10 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Hours | 3.0000 [2.000 to 4.000]

46. Primary Outcome: Apparent Terminal Half-life (T1/2) of GSK3439171A Following Single Dose-Part A (GSK3439171A 5 mg Only)
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36 and 48 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: GSK3439171A 5 mg
Number analyzed (Participants) | 6
Hours | 9.847 (46.4)

47. Primary Outcome: T1/2 of GSK3439171A Following Single Dose-Part A (GSK3439171A 10 mg, 30 mg, 60 mg, 120 mg and 180 mg)
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg
Number analyzed (Participants) | 6 | 5 | 6 | 6 | 6
Hours | 11.233 (44.6) | 11.956 (7.5) | 11.183 (17.8) | 11.761 (19.3) | 11.076 (22.1)

48. Primary Outcome: T1/2 of GSK3439171A Following Single Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 9
Hours | 15.348 (26.6) | 14.275 (32.4)

49. Primary Outcome: T1/2 of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: Day 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 7
Hours | 13.253 (23.8) | 11.584 (11.3)

50. Primary Outcome: T1/2 of GSK3439171A Following Single Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Hours | 11.908 (18.9)

51. Primary Outcome: T1/2 of GSK3439171A Following Repeat Dose-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: Day 10 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Hours | 10.948 (18.4)

52. Secondary Outcome: AUC(0 to t) of GSK3439171A (Food Effect)-Part C
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Hours*nanograms per milliliter | 16263.2 (27.0) | 14770.1 (29.0)
Statistical Analysis 1: Comparison: Part C: GSK3439171A 60 mg Fasted vs Part C: GSK3439171A 60 mg Fed; Test type: Other; Ratio = 0.93, 90% CI 2-sided [0.84 to 1.03] — Analysis was performed using Mixed Effect Model with treatment and period as fixed effect and participant as random effect. "Variance Components" covariance structure was used

53. Secondary Outcome: AUC(0 to Inf) of GSK3439171A (Food Effect)-Part C
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Hours*nanograms per milliliter | 16458.9 (27.4) | 14995.0 (29.7)
Statistical Analysis 1: Comparison: Part C: GSK3439171A 60 mg Fasted vs Part C: GSK3439171A 60 mg Fed; Test type: Other; Ratio = 0.93, 90% CI 2-sided [0.84 to 1.04] — [estimate comment as in outcome 52, analysis 1]

54. Secondary Outcome: Cmax for GSK3439171A (Food Effect)-Part C
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Nanograms per milliliter | 1155.60 (16.3) | 1025.45 (21.2)
Statistical Analysis 1: Comparison: Part C: GSK3439171A 60 mg Fasted vs Part C: GSK3439171A 60 mg Fed; Test type: Other; Ratio = 0.89, 90% CI 2-sided [0.79 to 1.01] — [estimate comment as in outcome 52, analysis 1]

55. Secondary Outcome: Tmax for GSK3439171A-Part C
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Hours | 3.0000 [1.000 to 4.033] | 4.0000 [1.500 to 4.017]

56. Secondary Outcome: T1/2 for GSK3439171A-Part C
Description: as for outcome 22
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
Number analyzed (Participants) | 11 | 11
Hours | 10.820 (13.7) | 11.679 (19.7)

57. Secondary Outcome: Dose Proportionality of GSK3439171A Using AUC(0 to t) Following a Single Dose-Part A
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Dose proportionality was assessed using Power model with fixed effects of logarithm of treatment and participant as random effect. Slope and 90% confidence interval for the slope are presented.
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- GSK3439171A 5 mg to 180 mg: Participants were administered single oral doses of GSK3439171A 5 mg, 10 mg, 30 mg, 60 mg, 120 mg and 180 mg in either treatment period 1, 2 or 3.
Arm/Group | GSK3439171A 5 mg to 180 mg
Number analyzed (Participants) | 18
Slope of log dose | 1.068 [1.001 to 1.136]

58. Secondary Outcome: Dose Proportionality of GSK3439171A Using AUC(0 to Inf) Following a Single Dose-Part A
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Dose proportionality was assessed using Power model with fixed effects of logarithm of treatment and participant as random effect. Slope and 90 % confidence interval for the slope are presented.
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3439171A 5 mg to 180 mg
Number analyzed (Participants) | 18
Slope of log dose | 1.057 [0.988 to 1.125]

59. Secondary Outcome: Dose Proportionality of GSK3439171A Using Cmax Following a Single Dose-Part A
Description: as for outcome 57
Time Frame: pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3439171A 5 mg to 180 mg
Number analyzed (Participants) | 18
Slope of log dose | 0.944 [0.892 to 0.997]

60. Secondary Outcome: Dose Proportionality of GSK3439171A Using AUC(0 to Tau) Following Repeat Dose-Part B
Description: as for outcome 57
Time Frame: Days 10 and 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- GSK3439171A 5 mg to 40 mg: Participants were administered once daily oral doses of GSK3439171A 5 mg, 11 mg and 40 mg for up to 14 days.
Arm/Group | GSK3439171A 5 mg to 40 mg
Number analyzed (Participants) | 25
Slope of log dose | 0.966 [0.863 to 1.069]

61. Secondary Outcome: Dose Proportionality of GSK3439171A Using Cmax Following Repeat Dose-Part B
Description: as for outcome 57
Time Frame: Days 10 and 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3439171A 5 mg to 40 mg
Number analyzed (Participants) | 25
Slope of log dose | 0.972 [0.877 to 1.066]

62. Secondary Outcome: Observed Accumulation Ratio for AUC (AUC[Ro])-Part B (GSK3439171A 5 mg and 11 mg)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. AUC(Ro) was calculated as Day17 AUC(0 to tau) divided by Day 1 AUC (0 to tau). Analysis was performed using Mixed effect model with AUC (0 to tau) as the response variable. Treatment, visit and treatment-by-visit interaction are added as fixed effects and participant as random effect. Ratio and 90% confidence interval of the ratio is presented.
Time Frame: Days 1 and 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 7
Ratio | 1.39 [1.29 to 1.49] | 1.52 [1.40 to 1.64]

63. Secondary Outcome: Observed Accumulation Ratio for AUC (AUC[Ro])-Part B (GSK3439171A 40 mg Only)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. AUC(Ro) was calculated as Day10 AUC(0 to tau) divided by Day 1 AUC (0 to tau). Analysis was performed using Mixed effect model with AUC (0 to tau) as the response variable. Treatment, visit and treatment-by-visit interaction are added as fixed effects and participant as random effect. Ratio and 90% confidence interval of the ratio is presented.
Time Frame: Days 1 and 10 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Ratio | 1.49 [1.39 to 1.60]

64. Secondary Outcome: Observed Accumulation Ratio for Cmax (RCmax)-Part B (GSK3439171A 5 mg and 11 mg)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. RCmax was calculated as Day17 Cmax divided by Day 1 Cmax. Analysis was performed using Mixed effect model with Cmax as the response variable. Treatment, visit and treatment-by-visit interaction are added as fixed effects and participant as random effect. Ratio and 90% confidence interval of the ratio is presented.
Time Frame: Days 1 and 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 7
Ratio | 1.18 [1.05 to 1.31] | 1.28 [1.13 to 1.45]

65. Secondary Outcome: Observed Accumulation Ratio for Cmax (RCmax)-Part B (GSK3439171A 40 mg Only)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. RCmax was calculated as Day10 Cmax divided by Day 1 Cmax. Analysis was performed using Mixed effect model with Cmax as the response variable. Treatment, visit and treatment-by-visit interaction are added as fixed effects and participant as random effect. Ratio and 90% confidence interval of the ratio is presented.
Time Frame: Days 1 and 10 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Ratio | 1.49 [1.33 to 1.66]

66. Secondary Outcome: Steady State Accumulation Ratio (Rss)-Part B (GSK3439171A 5 mg and 11 mg)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Rss was calculated as Day 17 AUC(0-tau) divided by Day 1 AUC(0-inf). Analysis was performed using Mixed Effect Model, with AUC(0-tau) and AUC(0-inf) as the response variables. Treatment, visit, parameter and parameter-by-treatment-by-visit interaction are added as fixed effects and participant as random effect. Ratio and 90% confidence interval of the ratio is presented.
Time Frame: Days 1 and 17 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 7
Ratio | 1.07 [1.01 to 1.14] | 1.21 [1.13 to 1.29]

67. Secondary Outcome: Steady State Accumulation Ratio (Rss)-Part B (GSK3439171A 40 mg Only)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. Pharmacokinetic parameters were calculated using standard non-compartmental analysis. Rss was calculated as Day 10 AUC(0-tau) divided by Day 1 AUC(0-inf). Analysis was performed using Mixed Effect Model, with AUC(0-tau) and AUC(0-inf) as the response variables. Treatment, visit, parameter and parameter-by-treatment-by-visit interaction are added as fixed effects and participant as random effect. Ratio and 90% confidence interval of the ratio is presented.
Time Frame: Days 1 and 10 (pre-dose, 0.083, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 60 and 72 hours post-dose)
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Ratio | 1.16 [1.10 to 1.23]

68. Secondary Outcome: Trough Plasma Concentrations at the End of Dosing Interval for Repeat Doses on Days 6, 7, 9, 10, 11, 15, 16 and 17-Part B (GSK3439171A 5 mg and 11 mg)
Description: as for outcome 22
Time Frame: pre-dose on Days 6, 7, 9, 10, 11, 15, 16 and 17
Population: Pharmacokinetic Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 9
Nanograms per milliliter
  pre-dose Day 6; n=9, 9 | 27.3206 (42.3) | 35.6842 (55.9)
  pre-dose Day 7; n=9, 9 | 29.5449 (44.5) | 41.6334 (61.5)
  pre-dose Day 9; n=9, 9 | 28.5910 (46.0) | 38.2703 (65.3)
  pre-dose Day 10; n=9, 9 | 29.2380 (44.1) | 35.4203 (76.8)
  pre-dose Day 11; n=9, 9 | 28.8443 (42.8) | 30.4420 (105.7)
  pre-dose Day 15; n=9, 9 | 26.2039 (58.0) | 30.8384 (247.3)
  pre-dose Day 16; n=9, 9 | 27.4434 (51.3) | 24.9684 (362.7)
  pre-dose Day 17; n=9, 7: number analyzed (Participants) | 9 | 7
  pre-dose Day 17; n=9, 7 | 28.5046 (47.3) | 48.0658 (52.9)

69. Secondary Outcome: Trough Plasma Concentrations at the End of Dosing Interval for Repeat Doses on Days 6, 7, 9 and 10-Part B (GSK3439171A 40 mg Only)
Description: as for outcome 22
Time Frame: pre-dose on Days 6, 7, 9 and 10
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Nanograms per milliliter
  pre-dose Day 6 | 184.1428 (40.4)
  pre-dose Day 7 | 209.1741 (37.8)
  pre-dose Day 9 | 211.2785 (37.0)
  pre-dose Day 10 | 215.1369 (36.9)

70. Secondary Outcome: Steady State Assessment Using Trough Plasma Concentration at the End of Dosing Interval for Repeat Dose-Part B (GSK3439171A 5 mg and 11 mg)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. The slope estimate of the day effect was obtained from Mixed Effect Model, with visit as the fixed effect and participant as random effect. The analysis was done separately for each treatment. "Variance Component" covariance structure was used. The back transformed slope and 90% confidence interval for the slope is presented.
Time Frame: pre-dose on Days 6, 7, 9, 10, 11, 15, 16 and 17
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Slope
Arm/Group | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg
Number analyzed (Participants) | 9 | 9
Slope | 1.000 [0.998 to 1.001] | 0.997 [0.994 to 1.001]

71. Secondary Outcome: Steady State Assessment Using Trough Plasma Concentration at the End of Dosing Interval for Repeat Dose-Part B (GSK3439171A 40 mg Only)
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis. The slope estimate of the day effect was obtained from Mixed Effect Model, with visit as the fixed effect and participant as random effect. The analysis was done separately for each treatment. "Variance Component" covariance structure is used. The back transformed slope and 90% confidence interval for the slope is presented.
Time Frame: pre-dose on Days 6, 7, 9 and 10
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Slope
Arm/Group | Part B: GSK3439171A 40 mg
Number analyzed (Participants) | 9
Slope | 1.003 [1.002 to 1.005]

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from the start of study treatment until Day 40 for Part A, until Day 34 for Part B and from start of study treatment until Day 29 for Part C.
Description: Non-SAEs and SAEs were collected in the Safety Population which comprised of all participants who took at least 1 dose of study intervention.
Arm/Group | Part A: Placebo | Part A: GSK3439171A 5 mg | Part A: GSK3439171A 10 mg | Part A: GSK3439171A 30 mg | Part A: GSK3439171A 60 mg | Part A: GSK3439171A 120 mg | Part A: GSK3439171A 180 mg | Part B: Placebo | Part B: GSK3439171A 5 mg | Part B: GSK3439171A 11 mg | Part B: GSK3439171A 40 mg | Part C: GSK3439171A 60 mg Fasted | Part C: GSK3439171A 60 mg Fed
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/9 | 0/9 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/9 | 0/9 | 0/9 | 0/9 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/17 | 0/6 | 2/6 | 2/5 | 2/6 | 1/6 | 1/6 | 4/9 | 5/9 | 8/9 | 3/9 | 1/11 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=17) | Part A: GSK3439171A 5 mg (N=6) | Part A: GSK3439171A 10 mg (N=6) | Part A: GSK3439171A 30 mg (N=5) | Part A: GSK3439171A 60 mg (N=6) | Part A: GSK3439171A 120 mg (N=6) | Part A: GSK3439171A 180 mg (N=6) | Part B: Placebo (N=9) | Part B: GSK3439171A 5 mg (N=9) | Part B: GSK3439171A 11 mg (N=9) | Part B: GSK3439171A 40 mg (N=9) | Part C: GSK3439171A 60 mg Fasted (N=11) | Part C: GSK3439171A 60 mg Fed (N=11)
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site laceration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 2 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site dermatitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT03627494/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT03627494/SAP_001.pdf